CLINICAL TRIAL: NCT03970993
Title: A Phase I/IIa Sporozoite Challenge Study to Assess the Safety, Immunogenicity and Protective Efficacy of Adjuvanted R21, Administered in Different Dose Schedules in Healthy UK Volunteers
Brief Title: VAC 072-An Efficacy Study of R21/MM in Different Dose Schedules
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC072
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Malaria
Keywords: Malaria challenge; Malaria vaccine
MeSH Terms: conditions — Malaria | interventions — 1-acetyl-1,2,3,3a,8,8a-hexahydro-8a-hydroxy-5-methoxypyrrolo(2,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Group 1a (Experimental): Volunteers will receive 3 doses of 10μg R21/50μg Matrix-M 4 weeks apart and an optional booster vaccination 12 months after the third dose
  Interventions: Biological: R21 Matrix-M vaccination; Biological: R21 Matrix-M vaccination booster
- Group 2a (Experimental): Volunteers will receive 3 doses of 10μg R21/50μg Matrix-M at 0, 4 and 24 weeks, followed by CHMI by sporozoite challenge (mosquito bite) 4 weeks later. If protected from malaria, volunteers will receive an optional booster vaccination 28 days prior to malaria rechallenge
  Interventions: Biological: R21 Matrix-M vaccination and CHMI; Biological: R21 Matrix-M vaccination booster
- Group 3a (Experimental): Volunteers will receive 3 doses of 10μg R21/50μg Matrix-M 4 weeks apart, followed by CHMI by sporozoite challenge (mosquito bite) 4 weeks later. If protected from malaria, volunteers will receive an optional booster vaccination 28 days prior to malaria rechallenge
  Interventions: Biological: R21 Matrix-M vaccination and CHMI; Biological: R21 Matrix-M vaccination booster
- Group 4a (Experimental): Volunteers will receive 2 doses of 50μg R21/50μg Matrix-M 4 weeks apart and a 3rd fractional dose of 10μg R21/50μg Matrix-M at 24 weeks. This is followed by optional CHMI by sporozoite challenge (mosquito bite) 4 weeks later
  Interventions: Biological: R21 Matrix-M vaccination and CHMI
- Group 5 (Experimental): Volunteers will receive 2 doses of 10μg R21/50μg Matrix-M 4 weeks apart and a 3rd fractional dose of 2μg R21/50μg Matrix-M at 24 weeks. This is followed by optional CHMI by sporozoite challenge (mosquito bite) 4 weeks later
  Interventions: Biological: R21 Matrix-M vaccination and CHMI
- Group 6 (No Intervention): They are infectivity control volunteers for the sporozoite challenge procedures: these volunteers are not vaccinated.
- Group 7 (No Intervention): They are infectivity control volunteers for the sporozoite challenge procedures: these volunteers are not vaccinated.
- Group 1b (Experimental): Volunteers will receive 3 doses of 10μg R21/50μg Matrix-M, 4 weeks apart followed by an optional vaccination booster 12 months after the third dose.
  Interventions: Biological: R21 Matrix-M vaccination; Biological: R21 Matrix-M vaccination booster
- Group 2b (Experimental): Volunteers will receive 3 doses of 10μg R21/50μg Matrix-M at 0, 4 and 24 weeks.
  Interventions: Biological: R21 Matrix-M vaccination
- Group 3b (Experimental): Volunteers will receive 3 doses of 10μg R21/50μg Matrix-M 4 weeks apart.
  Interventions: Biological: R21 Matrix-M vaccination
- Group 4b (Experimental): Volunteers will receive 2 doses of 50μg R21/50μg Matrix-M 4 weeks apart and a 3rd fractional dose of 10μg R21/50μg Matrix-M at 24 weeks.
  Interventions: Biological: R21 Matrix-M vaccination

INTERVENTIONS:
Biological: R21 Matrix-M vaccination — Three dose vaccination of 2μg, 10μg or 50μg of R21 and 50ug Matrix-M delivered intramuscularly
  Arms: Group 1a; Group 1b; Group 2b; Group 3b; Group 4b
Biological: R21 Matrix-M vaccination and CHMI — Three dose vaccination of 2μg, 10μg or 50μg of R21 and 50ug Matrix-M delivered intramuscularly. Volunteers then have the option to be challenged with malaria by mosquito bite
  Arms: Group 2a; Group 3a; Group 4a; Group 5
Biological: R21 Matrix-M vaccination booster — Optional R21 Matrix-M vaccination booster following a three dose vaccination schedule
  Arms: Group 1a; Group 1b; Group 2a; Group 3a

SUMMARY:
An open label, partially blinded clinical trial in which healthy volunteers will be administered experimental malaria vaccines. There will be seven experimental groups of volunteers, of which five receive vaccination with the novel malaria vaccine candidate, R21, in combination with the vaccine adjuvant, Matrix M.

The study will assess the safety & immune responses to vaccination, and the efficacy of the vaccine.

DETAILED DESCRIPTION:
Arms 1a & 1b receive vaccines at 3 vaccinations at 4 week intervals and a booster vaccination approximately 12 months after the first vaccination.

Arms 2a & 2b receive 3 vaccinations at 0, 4 and 24 weeks. The protected volunteers in 2a from the first malaria challenge, VAC072A, will receive a booster vaccination 28 days before the rechallenge, VAC072B.

Arms 3a and 3b receive 3 vaccinations at 0, 4 and 8 weeks. The protected volunteers in 3a from the first malaria challenge, VAC072A, will receive a booster vaccination 28 days before the rechallenge, VAC072B.

Arms 4a and 4b will receive 3 vaccinations at 0, 4 and 24 weeks. The third dose is fractional. Volunteers then have the option to be challenged 28 days after final vaccination.

Group 5 will receive 3 vaccinations at 0, 4 and 24 weeks. The third dose is fractional. Volunteers then have the option to be challenged 28 days after final vaccination.

Groups 6 & 7 are control groups and will receive controlled human malaria infection (CHMI)

Healthy volunteers will be recruited in England across four research sites in Oxford, London, and Southampton.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner.
* Women only: Must practice continuous effective contraception for the duration of the study.
* Agreement to refrain from blood donation during the course of the study.
* Agree to refrain from blood donation for at least 3 years after the end of their involvement in the study.*
* Written informed consent to participate in the trial.
* Reachable (24/7) by mobile phone during the period between CHMI and completion of antimalarial treatment.*
* Willingness to take a curative anti-malaria regimen following CHMI.*
* For volunteers not living close to the malaria challenge follow-up site (CCVTM, Oxford) agreement to stay in a hotel room close to the trial centre during a part of the study (from at least day 6.5 post mosquito bite until anti-malarial treatment is completed).*
* Answer all questions on the informed consent quiz correctly.*

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim- sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin)*
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data as assessed by the investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products) or malaria infection.
* Any history of anaphylaxis post vaccination.
* History of clinically significant contact dermatitis.
* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Pregnancy, lactation or intention to become pregnant during the study.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone*
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone*
* Any clinical condition known to prolong the QT interval and existing contraindication to the use of Malarone.*
* History of cardiac arrhythmia, including clinically relevant bradycardia and existing contraindication to the use of Malarone.*
* Clinically significant disturbances of electrolyte balance, eg, hypokalaemia or hypomagnesaemia
* Family history of congenital QT prolongation or sudden death and existing contraindication to the use of Malarone.*
* Contraindications to the use of both Riamet and Malarone*
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 25 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* Positive family history in both 1st and 2nd degree relatives < 50 years old for cardiac disease.*
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested. Procedures for identifying laboratory values meeting exclusion criteria are shown in Appendix A.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

  * Not applicable for volunteers who do not undergo CHMI (Groups 1, 4 and 5)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of adjuvanted R21 using different immunisation schedules in healthy malaria naïve volunteers | Solicited AEs will be collected for 7 days and Unsolicited AEs will be collected for 28 days. SAEs will be collected from enrolment until the end of the follow-up period
  Occurrence of solicited and unsolicited local and systemic adverse events
The efficacy (prevention of occurrence of P. falciparum parasitemia) of adjuvanted R21 against malaria sporozoite challenge, in healthy malaria-naïve volunteers using two immunisation regimes | Weeks 2 & 3 following malaria infection
  Assessed by PCR of adjuvanted R21 in two different vaccination regimes

SECONDARY OUTCOMES:
To assess humoral immunogenicity generated in malaria-naïve individuals by adjuvanted R21 using different immunisation schedules in healthy malaria-naïve volunteers. | Blood samples will be taken to assess immune responses at specified time points over the duration of the study
  To document immunogenicity measures, capturing humoral and cellular immune responses to R21 as follows: Anti-CS antibody titers
To assess the safety and tolerability of adjuvanted R21 using different immunisation schedules in healthy malaria-naïve volunteers following booster vaccination | Solicited AEs will be collected for 7 days and Unsolicited AEs will be collected for 28 days. SAEs will be collected from enrolment until the end of the follow-up period
  Occurrence of solicited and unsolicited local and systemic adverse events
To assess the efficacy of adjuvanted R21 against malaria sporozoite challenge in healthy malaria-naïve volunteers following a booster vaccination. | Week 2 following malaria infection
  To assess the efficacy (prevention of occurrence of P. falciparum parasitemia, assessed by PCR) of adjuvanted R21 against malaria sporozoite challenge, in healthy malaria-naïve volunteers following a booster vaccination.
To further assess the efficacy using different thresholds of adjuvanted R21 in two different vaccination regimes and compared to R21c against malaria sporozoite challenge, in healthy malaria-naïve volunteers. | Weeks 2 & 3 following malaria infection
  To further assess the efficacy using different thresholds, measured as time to P. falciparum parasitemia, assessed by PCR of adjuvanted R21 in two different vaccination regimes and compared to R21c against malaria sporozoite challenge, in healthy malaria-naïve volunteers.

OTHER OUTCOMES:
To evaluate further exploratory immunological end points in the vaccinees. | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, DPhill FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom
Locations (4):
- United Kingdom (4):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - CCVTM, University of Oxford, Churchill Hospital, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southampton